CLINICAL TRIAL: NCT02967146
Title: Anti-adhesive Effect and Safety of a Mixed Solid of Poloxamer, Gelatin and Chitosan(Mediclore®) After Axillary Dissection for Breast Cancer A Multicenter Double-blinded, Randomized Study
Brief Title: Anti-adhesive Effect and Safety of a Mixed Solid of Poloxamer, Gelatin and Chitosan(Mediclore®) After Axillary Dissection for Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seok Won Kim, MD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-08-194-002
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Breastcancer; Surgery: Axillary Dissection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Mediclore (Experimental)
  Interventions: Device: adhesive barrier
- Not done (No Intervention): Standard treatment for surgery

INTERVENTIONS:
Device: adhesive barrier — After having axillary dissection, investigator has to inject the mediclore on op site directly and suture the site.
  Arms: Mediclore

SUMMARY:
Anti-adhesive effect and Safety of a mixed solid of poloxamer, gelatin and chitosan(Mediclore®) after axillary dissection for breast cancer

DETAILED DESCRIPTION:
A Multicenter Double-blinded, Randomized Study

ELIGIBILITY:
Inclusion Criteria:

* the patients needed axillary dissection in breast cancer
* Written informed consent
* Patients without clinically significant lab
* the patients who are diagnosed 'positive for metastasis' by sentinel lymph node biopsy

Exclusion Criteria:

* having enrolled another clinical trials within 1 month
* Immunosuppression or autoimmune disease
* Anticoagulant, general steroids within a week from surgery
* Incompatible medications
* Serious diseases (heart failure, renal failure, liver failure, uncontrolled hypertension, diabetes mellitus, coagulation deficiencies)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
sum of ROM(range of motion) | 4weeks
  to compare the differences of sum of ROM between two groups comparision of the differences of sum of ROM between two groups ROM: forward flexion and horizontal abduction

SECONDARY OUTCOMES:
sum of ROM(range of motion) | 24weeks
  comparision of the differences of sum of ROM between two groups ROM: forward flexion and horizontal abduction
pain assessment (numeric pain rating scale) | 4weeks, 24weeks
  to compare the differences of the pain related with motions of upper limbs
Scoring DASH(Disablities of the arm, shoulder and hand) | 4weeks, 24weeks
  to compare the differences of the DASH score

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi HJ, Ryu JM, Chae BJ, Kim EK, Min JW, Shin HJ, Nam SJ, Yu J, Lee JE, Lee SK, Kim SW. Effect of Poloxamer-Based Thermo-Sensitive Sol-Gel Agent on Upper Limb Dysfunction after Axillary Lymph Node Dissection: A Double-Blind Randomized Clinical Trial. J Breast Cancer. 2021 Aug;24(4):367-376. doi: 10.4048/jbc.2021.24.e30. Epub 2021 Jun 17. PMID 34352935